## Dissemination and Implementation of a Videoconference Antimicrobial Stewardship Team (VAST)

ClinicalTrials.gov ID: NCT05319561

ICF document date: 03/20/2023 & 09/21/2021

Dear [NAME],

We are reaching out to you to ask for your participation in a research study. This study has been approved by VA Central Institutional Review Board. Drs. Jump and Evans are conducting research on the Videoconference Antimicrobial Stewardship Team (VAST).

A survey link has been attached to this email. The survey should take no longer than 20 minutes to complete.

Completion of the survey will indicate your willingness to participate in this research study. The decision to participate in this study is completely voluntary on your part. Refusal to take part in the study will involve no penalty. You may discontinue taking part at any time without any penalty.

The results of the survey will not be shared with colleagues, supervisors, or administrators. Only aggregate data will be shared with anyone outside of the research team.

[LINK]

Sincerely,

Drs. Jump and Evans

For additional information, please contact us at:

Robin Jump, MD, PhD: Charlesnika T. Evans, PhD, MPH:

## **Providers**

Greetings,

Our team is working on a VA Central IRB approved study to better understand the effectiveness of the Videoconference Antimicrobial Stewardship Team (VAST), in which you have been participating.

We are inviting you to participate in an interview to better understand your views as a member of the VAST.

This interview is not part of any performance measure. Your participation is voluntary. All data collected will be kept confidential and anonymous, findings will be aggregated and de-identified prior to reporting and neither you nor your site will be identified in any reports or publications.

We will ask for your permission to record the interview to assist our team during analysis. The audio recording and any notes generated will be stored on a secure VA drive accessible only by the project team. You may decide not to participate in the interview or to be recorded at any time.

Please let us know if you are willing to participate and we will work to schedule an interview time that is convenient for your schedule.

We appreciate your time and assistance in this effort.